CLINICAL TRIAL: NCT02345304
Title: A Study to Investigate the Effects of BI 1181181 on the Pharmacokinetics of Midazolam, Warfarin, Omeprazole and Digoxin in Healthy Male Subjects
Brief Title: Effect of BI 1181181 on Midazolam, Warfarin, Omeprazole and Digoxin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1344.3; 2014-004329-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
MeSH Terms: interventions — Omeprazole; Warfarin; Midazolam; Digoxin

ARMS (5):
- Treatment 3 (Experimental): single dose of midazolam + BI drug
  Interventions: Drug: Midazolam; Drug: BI 1181181
- Treatment 4 (Experimental): single dose of probe drugs + BI drug
  Interventions: Drug: Omeprazole; Drug: Midazolam; Drug: BI 1181181; Drug: Warfarin
- Treatment 5 (Experimental): single dose of digoxin + BI drug
  Interventions: Drug: BI 1181181; Drug: Digoxin
- Treatment 1 (Experimental): single doses of probe drugs
  Interventions: Drug: Warfarin; Drug: Omeprazole; Drug: Midazolam
- Treatment 2 (Experimental): single dose of digoxin
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Omeprazole
  Arms: Treatment 4
Drug: Warfarin
  Arms: Treatment 1
Drug: BI 1181181
  Arms: Treatment 5
Drug: Midazolam
  Arms: Treatment 4
Drug: Omeprazole
  Arms: Treatment 1
Drug: BI 1181181
  Arms: Treatment 4
Drug: Midazolam
  Arms: Treatment 3
Drug: Midazolam
  Arms: Treatment 1
Drug: Warfarin
  Arms: Treatment 4
Drug: BI 1181181
  Arms: Treatment 3
Drug: Digoxin
  Arms: Treatment 5
Drug: Digoxin
  Arms: Treatment 2

SUMMARY:
To assess the influence of different dose strengths of BI 1181181 on single dose kinetics of midazolam (CYP3A4 probe drug), warfarin (CYP2C9 probe drug), omeprazole (CYP2C19 probe drug) and digoxin (P-gp probe drug)

ELIGIBILITY:
Inclusion criteria:

* healthy male subjects
* age of 18 to 50 years
* body mass index (BMI) of 18.5 to 29.9 kg/m2
* Subjects must be able to understand and comply with study requirements

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) of midazolam and omeprazol after each dosing | up to 24 hours
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) of digoxin after each dosing | up to 96 hours
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) of warfarin after each dosing | up to 120 hours
Cmax (Maximum measured concentration the analyte in plasma) of midazolam and omeprazol after each dosing | up to 24 hours
Cmax (Maximum measured concentration the analyte in plasma) of digoxin after each dosing | up to 96 hours
Cmax (Maximum measured concentration the analyte in plasma) of warfarin after each dosing | up to 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1344.3.1 Boehringer Ingelheim Investigational Site, Biberach, Germany